CLINICAL TRIAL: NCT06771375
Title: Eye Movement Desensitization and Reprocessing (EMDR) to Treat Chronic Pruritus in a Multidisciplinary Tertiary Care Setting- a Feasibility Study
Brief Title: Eye Movement Desensitization and Reprocessing (EMDR) to Treat Chronic Pruritus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-02597, th24schaefert
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pruritus
Keywords: Eye Movement Desensitization and Reprocessing
MeSH Terms: interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: non-randomized, open-label two-arm pre-post design feasibility-study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): EMDR (Eye Movement Desensitization and Reprocessing)-Treatment of patients suffering from CP + Treatment as Usual (TAU).
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing
- Standard of care group (No Intervention): Treatment as Usual (TAU) - depending on the underlying disease

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing — EMDR is a psychotherapeutic approach originally designed for individuals suffering from trauma and post-traumatic stress disorder (PTSD). It facilitates the processing of memories through a structured eight-phase treatment, involving the patient's focused attention on traumatic images, thoughts, and sensations while simultaneously engaging in bilateral stimulation, typically through guided eye movements. This process aims to reduce the emotional distress associated with aversive memories, promoting adaptive coping mechanisms and psychological healing. Recently, the indications for the method have been extended so that EMDR is also used for chronic pain and depressive disorders.
  Arms: Intervention Group

SUMMARY:
Pruritus is a common symptom of numerous dermatological and non-dermatological conditions. Current treatments for chronic pruritus (CP) are often not fully effective and may have burdensome side effects. Recently, the trauma exposure technique Eye Movement Desensitization and Reprocessing (EMDR) that is recommended as first line treatment for posttraumatic stress disorder has been reported to be also effective in the treatment of CP in anecdotal clinical case observations. However, to the best of the investigator's knowledge, the efficacy of EMDR in CP has not yet been systematically explored. This study aims at addressing this unmet need in a prospective pilot study comparing EMDR versus treatment as usual (TAU).

ELIGIBILITY:
Inclusion Criteria:

* Provided written informed consent
* Age 18 to 75 years
* Skindex-29 (questionnaire) symptoms subscale ≥42
* Confirmed diagnosis CP
* Itch intensity of min. ≥ 4 on the 0-10 numerical rating scale within the last 7 days
* Stable course of treatment in the two weeks prior to the study

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g. due to language problems, severe psychiatric disorders such as delusional disorder, suicidality or dementia.
* Patients on phototherapy
* Acute attacks of an autoimmune disease such as Crohn's disease
* Serious cardiac disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Adherence (%) | up to 8 month
  Adherence/ receipt of intervention and retention will be assessed by tracking % of sessions completed, number of dropouts and number of patients completing final assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Chrysovalandis Schwale, Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No